CLINICAL TRIAL: NCT06901362
Title: Seroprevalence and Vaccination Rate of Hepatitis B Virus and Varicella-zoster Virus Among Medical Students Under Immunizing Program
Status: Completed | Type: Observational
Sponsor: Thammasat University (Other)
Collaborators: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Other Study IDs: MTU-EC-SA-0-159/67
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Healthy Adult
Keywords: hepatitis B virus; varicella-zoster virus; vaccination; immunizing program; medical students
MeSH Terms: conditions — Hepatitis B; Chickenpox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for measuring immunity levels against the hepatitis B virus and varicella-zoster virus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical students: Medical students aged 18 years or older

SUMMARY:
This study is a cross-sectional study. The study aims to determine the levels of immunity against hepatitis B virus and varicella-zoster virus in medical students.

DETAILED DESCRIPTION:
This study is a cross-sectional study aimed at determining the levels of immunity against the hepatitis B virus and varicella virus in medical students. Additionally, it aims to compare the rate of increase in immunity levels before and after receiving the hepatitis B and varicella-zoster vaccines in medical students. Medical students aged 18 years or older are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Medical students
* Age 18 years or older

Exclusion Criteria:

* Known cases of hepatitis B virus infection
* Known cases of varicella-zoster virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical students aged 18 years or older are included.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
The seroprevalence of hepatitis B virus | From enrollment to the end of treatment at 6 months
  The immunity level against the hepatitis B virus is assessed.
The seroprevalence of varicella-zoster virus | From enrollment to the end of treatment at 6 months
  The immunity level against varicella-zoster virus is assessed.

SECONDARY OUTCOMES:
The vaccination rate of hepatitis B virus | From enrollment to the end of treatment at 6 months
  The vaccination rate of hepatitis B virus is assessed.
The vaccination rate of varicella-zoster virus | From enrollment to the end of treatment at 6 months
  The vaccination rate of varicella-zoster virus is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, MD, Principal Investigator — Thammasat University Faculty of Medicine
Locations (1):
- Narongkorn Saiphoklang, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and documents will be available for sharing immediately after publication for a period of 2 years.
Access Criteria: All researchers will be able to access the IPD and supporting information via the repository website without restriction.

REFERENCES:
- [Result] Techasathit W, Ratanasuwan W, Sonjai A, Sangsiriwut K, Anekthananon T, Suwanagool S. Vaccination against hepatitis B virus: are Thai medical students sufficiently protected? J Med Assoc Thai. 2005 Mar;88(3):329-34. PMID 15962639
- [Result] Baer G, Bonhoeffer J, Schaad UB, Heininger U. Seroprevalence and immunization history of selected vaccine preventable diseases in medical students. Vaccine. 2005 Mar 14;23(16):2016-20. doi: 10.1016/j.vaccine.2004.03.073. PMID 15734076
- [Result] Balbi O, Baldi S, Rizza S, Pietroiusti A, Perrone S, Coppeta L. Seroprevalence survey for Varicella among healthcare workers and medical students in Italy. Hum Vaccin Immunother. 2021 Feb 1;17(2):372-376. doi: 10.1080/21645515.2020.1771989. Epub 2020 Jul 9. PMID 32643520
- [Result] Pourakbari B, Shahbaznezhad L, Parvaneh N, Nikkhah S, Mahmoudi S, Teymuri M, Alyari A, Mamishi S. Seroepidemiology of Varicella Zoster Virus among children, adolescents and medical students in a referral children medical center, Tehran, Iran. Iran J Microbiol. 2012 Sep;4(3):136-8. PMID 23066488
- [Result] Sheek-Hussein M, Hashmey R, Alsuwaidi AR, Al Maskari F, Amiri L, Souid AK. Seroprevalence of measles, mumps, rubella, varicella-zoster and hepatitis A-C in Emirati medical students. BMC Public Health. 2012 Dec 5;12:1047. doi: 10.1186/1471-2458-12-1047. PMID 23217121
- [Result] Cardenas-Perea ME, Gomez-Conde E, Santos-Lopez G, Perez-Contreras I, Diaz-Orea MA, Gandara-Ramirez JL, Cruz Y Lopez OR, Marquez-Dominguez L, Sosa-Jurado F. Hepatitis B surface antibodies in medical students from a public university in Puebla, Mexico. Hum Vaccin Immunother. 2016 Jul 2;12(7):1857-62. doi: 10.1080/21645515.2016.1151587. Epub 2016 May 12. PMID 27171749
- [Result] Sartorelli P, Occhialini F, Miceli R, Pietronigro A, Bianciardi L, Salini C, Messina G. The seroprevalence of the hepatitis B virus in Italian medical students after 3 decades since the introduction of universal vaccination. Int J Occup Med Environ Health. 2022 Feb 15;35(1):75-80. doi: 10.13075/ijomeh.1896.01835. Epub 2021 Aug 25. PMID 34448470
- [Result] Tesfa T, Hawulte B, Tolera A, Abate D. Hepatitis B virus infection and associated risk factors among medical students in eastern Ethiopia. PLoS One. 2021 Feb 19;16(2):e0247267. doi: 10.1371/journal.pone.0247267. eCollection 2021. PMID 33606777
- [Result] Rathi A, Kumar V, Majhi J, Jain S, Lal P, Singh S. Assessment of knowledge, attitude, and practices toward prevention of hepatitis B infection among medical students in a high-risk setting of a newly established medical institution. J Lab Physicians. 2018 Oct-Dec;10(4):374-379. doi: 10.4103/JLP.JLP_93_18. PMID 30498306
- [Result] Yoda T, Katsuyama H. Analysis of antibody-negative medical students after hepatitis B vaccination in Japan. Hum Vaccin Immunother. 2021 Mar 4;17(3):852-856. doi: 10.1080/21645515.2020.1788309. Epub 2020 Aug 5. PMID 32755433
- [Result] Bianchi FP, Tafuri S, Larocca AMV, Germinario CA, Stefanizzi P. Long -term persistence of antibodies against varicella in fully immunized healthcare workers: an Italian retrospective cohort study. BMC Infect Dis. 2021 May 25;21(1):475. doi: 10.1186/s12879-021-06180-x. PMID 34034659
- [Result] Phattraprayoon N, Kakheaw J, Soonklang K, Cheirsilpa K, Ungtrakul T, Auewarakul C, Mahanonda N. Duration of Hepatitis B Vaccine-Induced Protection among Medical Students and Healthcare Workers following Primary Vaccination in Infancy and Rate of Immunity Decline. Vaccines (Basel). 2022 Feb 10;10(2):267. doi: 10.3390/vaccines10020267. PMID 35214725